CLINICAL TRIAL: NCT05103488
Title: Effectiveness of Comprehensive Palliative Care on Improving Quality of Life and Psychological Distress Among Cancer Patients in Vietnam - a Randomized Control Trial
Brief Title: Comprehensive Palliative Care for Cancer Patients in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam Palliative Health Care Society (Other)
Collaborators: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PC-MDT
Record Dates: First submitted 2021-10-02; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Advanced Cancer; Psychological Distress; Quality of Life
Keywords: holistic palliative care; supportive care; psychosocial support; interdisciplinary approach; social work; palliative care; advanced cancer; quality of life; Vietnam
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Comprehensive palliative care (CPC) is multidisciplinary inpatient care that aims to respond to patients' suffering in many aspects: physical, psychological, social, and spiritual. It is basically a standard palliative care service in Vietnam with additional psychosocial and spiritual support with a multidisciplinary approach. CPC is provided by seven doctors, 20 nurses, two social workers, a pharmacist, and a psychologist. CPC could go parallel with oncology care or be the primary care for patients.
  The psychosocial and spiritual supports are mainly provided by social workers. Psychologist and religious will get involved when patient need advance care. The psychosocial intervention is individualized for each patient based on their individual situation, issues, and decision.
  Interventions: Other: Comprehensive palliative care
- Control (Other): Patients who are randomized to the control group will receive the standard palliative care in Vietnam. They can assess to the same palliative care for their physical symptoms as patients in the intervention group do. They can also access psychosocial and spiritual support from the resources that available for them before entering to the study. If they request for social or financial support, their care team can reach out to the social work departments. Patients who are in need can receive mental health care from psychiatrists from the psychiatrist unit at UMC.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Comprehensive palliative care — CPC is multidisciplinary inpatient care that aims to respond to patients' suffering in many aspects: physical, psychological, social, and spiritual. It is basically a standard palliative care service in Vietnam with additional psychosocial and spiritual support with a multidisciplinary approach.
  Arms: Intervention
Other: Standard of care — Patients who are randomized to the control group will receive the standard palliative care in Vietnam. They can assess to the same palliative care for their physical symptoms as patients in the intervention group do. They can also access psychosocial and spiritual support from the resources that available for them before entering to the study. If they request for social or financial support, their care team can reach out to the social work departments. Patients who are in need can receive mental health care from psychiatrists from the psychiatrist unit at UMC.
  Arms: Control

SUMMARY:
There are exponential increases in cancer incidence and mortality worldwide and in Vietnam. Cancer affects patient's quality of life, which can be improved by palliative care. In Vietnam, due to a shortage in human resources for social workers, palliative care is mainly focused on medical aspect. A new comprehensive palliative care model, that provides multidisciplinary support including psychosocial support to patients, was developed. This research's objective is to evaluate the effectiveness of comprehensive palliative care (CPC) on improving the quality of life among cancer patients at a hospital in Vietnam.

This randomized control trial is performed among 100 advanced cancer patients at University Medical Center at Ho Chi Minh city, Vietnam.The measurement tools include the Vietnamese Palliative Care Outcome Scale (VietPOS), the 5-level EQ-5D (EQ-5D-5L), Hospital Anxiety and Depression Scale (HADS) and Zarit Burden Interview (ZBI). Data collection has been conducting through face-to-face interviews three times: baseline, week 3, and week 6. Paired t-test (or Wilcoxon Rank sum test) and Student-t-test (or Mann -Whitney U test) will be used to evaluate and compare changes in quality of life and psychological distress within and between groups. Intention- to - treat analysis is used in the study.

This is the first research that study the effectiveness of a palliative care psychosocial intervention on cancer patients in Vietnam. The result can be used to advocate for multidisciplinary palliative care in Vietnam.

DETAILED DESCRIPTION:
Background Vietnam, a Southeast Asian country with a population of 97 million, is still facing both communicable and non-communicable conditions, in which cancer is on the rise. In a report by GLOBOCAN 2020, the number of new cancer cases were 182,563 cases with around 122,690 cancer deaths in 2020 (World Health Organization, 2020). Living and dying with cancer, patients not only cope with their long-term physical conditions but also deal with complex sufferings which significantly affect their quality of life (Arman, Rehnsfeldt et al, 2004; Cherny et al, 1994; Hui et al, 2015). Cancer patients suffer from clusters of symptoms from physical, psychosocial issues as pain (35-96%), anorexia (30-92%), depression (3-77%) (Solano, et al, 2006). A recent Vietnamese study in stage III and IV cancer patients found out that health related quality of life and general health were reported as bad and very bad in about 23% and 52% of patients, respectively. (Huyen et al., 2021) Palliative care is one of the essential components in cancer programs, along with prevention, early detection, diagnosis, and treatment to reduce the incidence, mortality from cancer, and improve the quality of life for cancer patients. (WHO, 2002). In 2006, Vietnam's MoH endorsed the very first national guideline for provision of palliative care in Vietnam (Krakauer et al., 2018). The traditional palliative care team in Vietnam consists of two main components of physician and nurse (Krakauer et al., 2018). However, surveys among those palliative care clinicians revealed that they felt more competent providing physical care than psychological, social, and spiritual care (Nguyen et al., 2014; Tsao et al., 2019) To further promote the role of social work in hospitals, the Vietnamese MoH issued Circular 43/2015/TT-BYT regulation on the required tasks and organizations of social work in hospital settings. Evidence of efficacy from palliative care social support provided by social workers is needed to advocate for more allocation of resources.

Aims and objectives The aim of this study is to evaluate the effectiveness of a multidisciplinary CPC on improving quality of life and psychological distress among advanced cancer patients at University Medical Center in Vietnam.

The first objective is to assess the effect of the multidisciplinary CPC on cancer patient's quality of life. The second objective is to assess the effect of the multidisciplinary CPC on cancer patient's psychological distress.

Methods/Design Setting CPC is an inpatient hospital based in the Palliative and Geriatrics Unit at the University of Medical Center in Ho Chi Minh city. Each year, it serves more than 2 million outpatients per day (approximately 7000 patients/day); 55,000 inpatients. The unit has 30 fixed bed capacity but could mobilize up to 20 beds from other wards when needed. The area has very limited resources for home-based palliative care and community services for hospice.

Recruitment procedure Participants are recruited among cancer patients referred to palliative care. The research coordinator sends the trial's information and an invitation to eligible patients, and to get the consent form.

Randomization and blinding Block randomization. Before the first participant enrolled, a researcher created a block randomization list (block size = 4) by using Sealed Envelope (Sealed Envelope Ltd, 2020). Each week, an independent research coordinator not involved in the treatment assigned patients who finished their consent forms into groups based on the order of the list. The study is an open-label study due to the type of intervention.

Data collection. Data was collected through face-to-face interviews by 5 nurses who were not in patients' care team. Training was provided to all the data collectors to reduced bias and ensure quality of the data. It is required to conduct the questionnaire with a reasonable amount of time that did not exhaust patients. The interview schedule was arranged by the trial coordinator, then email to the interviewers. Data was collected as soon as a patient enrolled to the study. Then data collection was repeated at 3rd week and 6th week.

Intervention arm CPC is multidisciplinary inpatient care that aims to respond to patients' suffering in many aspects: physical, psychological, social, and spiritual. It is basically a standard palliative care service in Vietnam with additional psychosocial and spiritual support with a multidisciplinary approach. CPC is provided by seven doctors, 20 nurses, two social workers, a pharmacist, and a psychologist. CPC could go parallel with oncology care or be the primary care for patients.

The clinical palliative care team in the CPC intervention is a comprehensive group of multidisciplinary professionals who share a common goal to help patients manage their life-limiting illnesses. The multidisciplinary team arrange a team meeting once a week to discuss all the cases. The team member will share their concerns and collaborate in care planning.

The psychosocial and spiritual supports are mainly provided by social workers. Psychologist and religious will get involved when patient need advance care. The psychosocial intervention is individualized for each patient based on their individual situation, issues, and decision. All assessments for patients' psychosocial and spiritual distresses were conducted in the first week after enrolling to CPC. Patients can be discharged in different time based on their treatment and health conditions. CPC intervention is continued after patients are discharge though telephone calls. Due to COVID pandemic, home visit is not appropriate.

Control arm Patients who are randomized to the control group will receive the standard palliative care in Vietnam. They can assess to the same palliative care for their physical symptoms as patients in the intervention group do. They can also access psychosocial and spiritual support from the resources that available for them before entering to the study. If they request for social or financial support, their care team can reach out to the social work departments. Patients who are in need can receive mental health care from psychiatrists from the psychiatrist unit at UMC.

Sample size calculation Based on a study by Margareta Brännström et al. (Brännström & Boman, 2014), we estimated that a sample size of at least 41 participants in each group was needed to detect a mean difference of 8.60 in EQ-5D-5L score with a standard deviation of 13.70, and at 5% significance level, power of 80%. Due to the advanced stage of illness in the patients we estimated an attrition rate of 20% which meant that at least 50 participants were needed in each group.

Analysis We described and compared baseline data between the intervention and the control group using parametric and non-parametric tests as appropriate. We used t-test to compare the primary outcome, change in EQ-5D-5L after six weeks, between groups. Analyses of secondary outcomes included comparing domain of VietPOS, psychological distress and caregiver burden between groups. We used multiple imputation to deal with missing data. The alpha level for all statistical analyses was set at two-sided 0.05. All analyses were performed using R software.

Ethics approval Ethics approval for the study was gained from the ethics committee of University Medical Center at Ho Chi Minh city (Ref. 33/GCN-HĐĐĐ), obtained on 15/07/2020. The study protocol is retrospectively registered with ClinicalTrials.gov (NCT01165034). The delayed registration was due to the lack of human resource and technical support during the COVID-19 epidemics in Ho Chi Minh city, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 70
* In their first week of hospitalization
* Diagnosed with stage 3 or 4 of any cancer.

Exclusion Criteria:

* Patients with HIV, current pregnancy, or cognitive problems
* Could not communicate,
* Could not speak Vietnamese,
* Could not provide informed consent and questionnaires.
* Currently receiving palliative care services from other medical institutions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change of Quality of Life From Baseline to Week 6 by assessing The 5-level EQ-5D (EQ5D-5L) | 6 weeks
  Primary outcome is the change of quality of life after assed by the change of the total score of the 5-level EQ-5D questionnaire. The 5-level EQ-5D version was introduced by the EuroQol Group in 2009. It comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems, some problems, severe problems and unable to do. Each level of answer consists of each level of score ranges from 1 to 5. Each participant will have a health status consisting of 5 digits. Using the set of weights from Vietnamese population provided from the EuroGroup, we can convert each EQ-5D health state into a single summary index value. The index value ranges from 0 to 1, higher scores meaning better health quality.

SECONDARY OUTCOMES:
Change of Symptom Burden From Baseline to Week 6 by assessing the Vietnamese Palliative Outcome Scale (VietPOS) | 6 weeks
  The Vietnamese version of Palliative Care Outcome Scale was adapted and validated from the African-Palliative Outcome Scale in an unpublished study by a multi-institution research team of Dr Pham Thi Van Anh, Dr Eric Krakauer and Dr Richard Harding, endorsed by Vietnam's MoH. The Vietnamese Palliative Outcome Scale consists of 16 items, involving 4 domains: physical symptoms, psychological symptoms, psychosocial concerns, and caregiver concerns. Answers are given on a 6-point Likert scale, except for item 10, which is an open question on main problems experienced by the patient. The score for each item ranges from 0 to 5. The scores are calculated separately for patient and caregiver. Patient's symptom burden is calculated by 14 items for patient, total maximum score of 70, with higher scores meaning more severe burden. Caregiver's symptom burden is calculated by 8 items for caregiver, total maximum score of 40, with higher scores meaning more severe burden.
Change of Psychological distress From Baseline to Week 6 using Hospital Anxiety and Depression Scale (HADS) | 6 weeks
  Depression and anxiety symptoms is assessed by the Vietnamese version of the Hospital Anxiety and Depression Score. The scores are reported separately for the Depression subscale and the Anxiety subscale. Depression on a 0-21 scale, with lower scores corresponding to lower depression and higher scores corresponding to higher depression. Anxiety on a 0-21 scale, with lower scores corresponding to lower anxiety and higher scores corresponding to higher anxiety
Change of Caregiver burden From Baseline to Week 4 by Zarit Burden Interview (ZBI) | 6 weeks
  Carer burden is assessed with Zarit Burden Interview. The tool was developed by Zarit Bédard et al. in 2001 to measure subjective burden among caregivers of adults with dementia. The 22-item self-report version with each question is scored on a 5-point Likert scale ranging from - never (score 0) to nearly always present (score of 4). Total scores range from 0 (low burden) to 88 (high burden) with higher score correlating with greater caregiver burden

CONTACTS AND LOCATIONS:
Overall Officials: Quynh Truong, SW, MPH, Principal Investigator — Vietnam Palliative Health Care Society
Locations (1):
- Vietnam Palliative Health Care Society, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No